CLINICAL TRIAL: NCT01168700
Title: A PROSPECTIVE, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL OF THE SUPPLEMENTATION WITH KIOLIC® IN PATIENTS WITH DIAGNOSIS OF METABOLIC SYNDROME TO IMPROVE ENDOTHELIAL FUNCTION AND INFLAMMATORY STATE. "KYMES"
Brief Title: Trial of Supplementation With Aged Garlic Extract to Improve Endothelial Function in Patients With Metabolic Syndrome
Acronym: Kymes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Santander (Other)
Collaborators: Instituto de Salud de Bucaramanga (Other)
Responsible Party: Patricio López-Jaramillo, Universidad de Santander
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kymes-Wakunaga-UDES
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome, Aged Garlic Extract, Insulin, inflammation, endothelium.
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Inflammation | interventions — kyolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 1.2 g per day for 12 weeks, followed by a second treatment period with aged garlic extract during 12 more weeks.
  Interventions: Drug: Placebo
- Aged garlic extract (Kyolic ®) (Experimental): Aged garlic extract, 1.2 g per day for 12 weeks, followed by a second treatment period with placebo during 12 more weeks.
  Interventions: Drug: aged garlic extract

INTERVENTIONS:
Drug: aged garlic extract — Aged garlic extract, 1.2 g per day for 12 weeks
  Other Names: Kyolic
  Arms: Aged garlic extract (Kyolic ®)
Drug: Placebo — Placebo 1.2 g per day for 12 weeks.
  Arms: Placebo

SUMMARY:
Many studies have addressed the relationship between metabolic syndrome and cardiovascular disease. Risk factors include abdominal obesity, insulin resistance, abnormal lipid profile and hypertension. It is proposed that this condition leads to an increase in the production of inflammatory substances and endothelial dysfunction.

New therapies have been studied to improve control of metabolic disorders and reduce the endothelium damage. Aged garlic extract (Kyolic®) is a promising intervention that has antithrombotic and antioxidant properties. At the moment there is not data about the effects of supplementation with AGE in the endothelial function of patients with metabolic syndrome. Thus, the purpose of this study is to investigate if the supplementation with Kyolic® can alter the plasma levels of inflammatory markers, insulin and the endothelial function of patients with metabolic syndrome.

Methods and design: A randomized, cross over, double-blind, placebo-controlled trial will be performed to assess the effects of 1.2 g of Kyolic in insulin resistance and endothelial function of 46 patients with diagnosis of metabolic syndrome. The participants will be recruited from the primary care centers from E.S.E ISABU Bucaramanga. All subjects who meet the inclusion criteria will be randomly assigned to two periods of 12 weeks (Kyolic and placebo). Control visits will be programmed monthly to verify compliance and the presence of adverse events. Outcome variables (endothelial function assessed by flow mediated vasodilation, inflammatory markers, insulin plasma levels) will be evaluated at the initial visit and after 12 and 24 weeks of treatment.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) have become the main cause of death worldwide. It is estimated that 3.8 million men and 3.4 million women die every year from this cause (WHO 2006). In addition, an increase of 47 to 83 million disability-adjusted life years (DALY) between 1990 and 2020 has been projected for this disease (WHO 2006b). It is calculated that 5.3 million deaths by CVD occur in developed countries, while 8 to 9 million deaths occur in developing countries (Yusuf et al 2001; Lopez 1993). In Colombia, the death rate for CHD in 20-84 year old subjects increased from 58.5 per 100.000 in 1980 to 103.2 in 1996. Only 30% of this increase could be attributed to population aging (Lopez-Jaramillo et al 2001). From 1997 to 2001 acute myocardial infarction (AMI), stroke and diabetes mellitus type 2 (DM 2) were responsible for 213.150 deaths (19.6%). Together, these deaths exceeded those due to violent causes, which for several years were the first cause of death in this country.

The INTERHEART study (Yusuf 2004) identified the risk factors associated with AMI in 52 developed and developing countries. Smoking, hypertension, abnormal lipids, abdominal obesity (AO), diabetes and psychosocial stress were associated with ischemic disease in all regions of the world with no differences in age and gender. However, Lanas et al. (2007) reported the results of 1237 Latin American subjects from Brazil, Argentina, Chile and Colombia, included in the INTERHEART study, demonstrated that central obesity was the most important risk factor associated with AMI in this population, much more than in the entire population of the study. We have proposed that the biological response to obesity in developed countries is different than in developing countries, and that this response is modulated through epigenetic regulation (Lopez-Jaramillo et al 2008).

The consumer society has given rise to an increase in the prevalence of overweight, obesity, hypertension, diabetes mellitus type 2 (DM2) and finally metabolic syndrome (MS). Changes in the nutritional and physical habits are the main characteristics involved in the fast economic transition, where the over nutrition and the increased consumption of saturated fat and cholesterol, low intakes of polyunsaturated fat and lower physical activity are common determinants (Pi-Sunyer 2002).

The metabolic syndrome is a set of risk factors for diabetes mellitus type 2 and cardiovascular disease, characterized by the presence of resistance to insulin and compensating hyperinsulinemia, associate to alterations of carbohydrates and lipids metabolism, elevated arterial blood pressure and obesity (Pineda 2008). In 1988, Reaven observed that several risk factors (dislipidemia, hypertension, hyperglycemia) tended to be together. This set was named syndrome X (Reaven 1988). The name metabolic syndrome like a diagnostic entity with defined criteria was introduced by the WHO in 1998 (Alberti, Zimmet 1998). The metabolic syndrome prevalence varies according to some factors such as gender, age, ethnic group, but it is located between 15% to a 40%, being greater in the population of hispanic origin (Ford et al 2002). Metabolic syndrome is important in Colombia, where the population have a major sensibility to the development of an atherogenic lipid profile (Perez et al 2003), and low grade inflammation correlated to lower levels of abdominal obesity have been described (Garcia et al 2007). These factors are associated with an increase of the vascular reactivity to the angiotensin II stimulus (Rueda-Clausen et al 2007), hormone that is also produced in the visceral adiposity (17). The latter, at the endothelial level, increases the TNF production (Arenas et al 2004), a proinflammatory citokine that stimulates the hepatic production of C reactive protein (CRP), which in our population in situations such as abdominal obesity in adults (Garcia et al 2007) and children (Lopez-Jaramillo 2008b), arterial hypertension (Rueda-Clausen et al 2007), endothelial dysfunction (Garcia et al 2007b) and pregnancy induced hypertension (Teran et al 2001) is presented in higher levels than in other populations.

Recent studies have shown that obesity, insulin resistance and diabetes type 2 are proinflammatory states (Grundy et al 2004). It has been demonstrated that enlargement of adipocytes is frequently observed in obesity and in pre-diabetic individuals and in type 2 diabetics (Lundgren et al 2007). The increased adipocyte size may represent a failure in the recruitment of new adipocytes due to impaired differentiation; it has recently been shown that fat cell enlargement is an independent marker of insulin resistance (Rotter et al 2003). Cell size expansion leads to a reduction in the production of anti-inflammatory adipokines (like adiponectin) while proinflammatory cytokines (like IL-6, and PCR) are markedly increased (Rotter et al 2003).

Recent therapies have been introduced to achieve a control of metabolic disorders and reduce the endothelium damage of the metabolic syndrome. The garlic (Allium sativum) has been shown to improve blood lipids (Zlatkis et al 1953; Chi 1982; Shoetan et al 1984; Gebhart 1991;Welch et al 1992; Gebhart 1993; Yeh, Yeh 1994;), to have antithrombotic effects (Srivastava, Tyagi 1993), to decrease antiplatelet aggregation (Kiesewetter et al 1993) and to have antioxidative properties, (Sendl et al 1992; Yamasaki et al 1993). Besides, it has been reported that garlic stimulates the phagocytotic function of macrophage and lymphocyte proliferation (Tadi et al 1990). These effects are produced largely due to its high content of organosulfur compounds and antioxidant activity. However fresh garlic may cause indigestion and its pungent odor that lingers on the breath and skin can be a social deterrent. These disagreeable effects of fresh garlic are due to allicin, an oxidant released upon cutting or chewing the clove.

An alternative source of garlic that is odorless and rich in antioxidants is aged garlic extract (AGE) (Amagase et al 2001; Borek 2001). The well-standardized and highly bioavailable supplement is produced by prolonged extraction and aging of organic fresh garlic at a stable room temperature. The process converts unstable compounds, such as allicin, to stable substances and produces high levels of water-soluble organosulfur compounds. These include S-allylcysteine (SAC), AGE's major component, and S-allylmercaptocysteine, unique to AGE. Among other compounds present are low amounts of oil-soluble organosulfur compounds, flavonoids, a phenol, allixin, selenium, and saponins.

AGE has demonstrated to be useful in the reduction of the arterial tension; Steiner et al (Steiner et al 1996) realized a double-blind crossover study comparing the effect of aged garlic extract with placebo on blood lipids in a group of 41 moderately hypercholesterolemic men. Their results show that there was a 5.5% decrease in systolic blood pressure and a modest reduction of diastolic blood pressure in response to aged garlic extract. Slowing et al (2001) found that intake of garlic can prevent diet-induced hypercholesterolemia and vascular alteration in the endothelium-dependent relaxation associated with atherosclerosis, Macan et al (2006) administered AGE or placebo at a dose of 5 mL twice a day for 12 wk. to patients whom also received warfarin for 12 weeks, after this period the levels of HDL in the garlic group was higher compared with the placebo group.

Most of the effects of age garlic extract (AGE) can be explain because its levels of antioxidant compounds, whom increases nitric oxide production and decreases the output of inflammatory cytokines, the latter has been demonstrated in cultured cells.

Nitric oxide (NO) is an important intercellular and intracellular messenger with a major role in controlling the physiological function of the cardiovascular system (Palmer et al 1987; Moncada et al 1991). It is synthesized from L-arginine by NO synthases (NOSs) in many of the cells of the cardiovascular system, including endothelial cells, macrophages, smooth muscle cells, platelets and fibroblasts (42). Three kinds of NOSs, neuronal constitutive NOS (ncNOS), inducible NOS (iNOS) and endothelial constitutive NOS (ecNOS), were reported to be responsible for NO biosynthesis in these cells (Kerwin et al 1995). NO derived from ecNOS was reported to modulate vasomotor tone, inhibition of platelet aggregation and adhesion, inhibition of leucocyte migration, suggesting that NO could explain the anti-atherogenicity actions of the vascular endothelium (Moncada et al 1991).

Flow-mediated dilation (FMD), a noninvasive method that uses high-resolution ultrasonography, is an established test to assess endothelial function. The FMD technique measures the changes in the brachial artery diameter as a response to shear stress, and it is partially dependent on the capacity of endothelial cells to release nitric oxide (Celermajer et al 1992). This method has been validated in Colombian population (Accini et al 2001; Lopez-Jaramillo et al 2004) and has been used to evaluated the effect of AGE in endothelial function. Williams et al (2005) conducted a trial in 15 men with angiographically proven coronary artery disease in a randomized, placebo-controlled, cross-over design with 2-week treatment and washout periods. During AGE supplementation, FMD increased significantly (p = 0.04) from the baseline (44%) and mainly in men with lower baseline FMD. Levels of FMD at the end of AGE treatment were significantly (p = 0.03) higher compared with the corresponding levels at the end of placebo treatment.

However, at the moment there is not data about the effect of supplementation with AGE in the endothelial function in patients with metabolic syndrome. Thus, the purpose of this study is to investigate if the supplementation of Kyolic® can alter the levels of inflammatory markers and the endothelial function (measured by VMF) in patient with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old with metabolic syndrome diagnosed by the presence of central obesity (waist circumference ≥ 90cm (male), ≥ 80 cm (female)) and two of the following criteria:
* Triglycerides ≥ 150 mg/dl
* High density lipoprotein cholesterol <40 mg/dL (male),<50 mg/dL (female)
* Blood pressure ≥ 130/85 mmHg
* Fasting plasma glucose ≥ 100 mg/dl

Exclusion Criteria:

* Garlic allergy
* Patients with psychiatric disorders that prevent proper decision-making
* Patients with infections or inflammatory conditions
* Presence of coronary artery disease
* Presence of severe chronic or terminal illnesses.
* Presence of diseases that compromise the immune system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Endothelial function assessed by flow mediated vasodilation and plasma levels of nitrites/nitrates | 12, 24 weeks
  The flow mediated vasodilation is a non-invasive diagnostic test using high-resolution doppler ultrasound, that measures the changes in diameter of the brachial artery in response to increased blood flow (reactive hyperemia).
  The plasma levels of nitrites/nitrates will be determined by immunoassay (R&D Systems, Inc)

SECONDARY OUTCOMES:
Plasma concentrations of C-reactive protein and interleukin-6 | 12, 24 weeks
  During the initial and follow-up visits, a blood sample will be taken to determine C-reactive protein by high sensitivity chemiluminescent immunometric assay (IMMULITE 1000, DPC, Los Angeles, CA) and Interleukin-6 by immunoassay (Biosource International, Camarillo, CA)
Plasma insulin and glucose levels | 12, 24 weeks
  Blood samples will be taken at the initial and follow-up visits (12,24 weeks) to determine blood glucose by automatic colorimetric method (Baker System 9120 AX, Biochem Immunosystem, Allentown, PA)and insulin plasma levels by high sensitivity chemiluminescent immunometric assay (IMMULITE 1000, DPC, Los Angeles, CA).
Waist and hip circumference | 12, 24 weeks
  Anthropometric measures will be determined at the initial and follow-up visits (12,24 weeks).
Plasma levels of Adiponectin | initial visit, 12, 24 weeks
  Blood samples will be taken at the initial and follow-up visits (12,24 weeks) to determine adiponectin by Human Adiponectin/Acrp30 Quantikine ELISA (R&D Systems, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio López-Jaramillo, MD, PhD, Principal Investigator — Universidad de Santander
Locations (1):
- Medicine School, Universidad de Santander, Bucaramanga, Santander Department, Colombia

REFERENCES:
- [Background] Yusuf S, Reddy S, Ounpuu S, Anand S. Global burden of cardiovascular diseases: part I: general considerations, the epidemiologic transition, risk factors, and impact of urbanization. Circulation. 2001 Nov 27;104(22):2746-53. doi: 10.1161/hc4601.099487. PMID 11723030
- [Background] Lopez AD. Assessing the burden of mortality from cardiovascular diseases. World Health Stat Q. 1993;46(2):91-6. PMID 8303909
- [Background] Lopez-Jaramillo P, Casas JP, Bautista L, Serrano NC, Morillo CA. An integrated proposal to explain the epidemic of cardiovascular disease in a developing country. From socioeconomic factors to free radicals. Cardiology. 2001;96(1):1-6. doi: 10.1159/000047379. PMID 11701934
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Lanas F, Avezum A, Bautista LE, Diaz R, Luna M, Islam S, Yusuf S; INTERHEART Investigators in Latin America. Risk factors for acute myocardial infarction in Latin America: the INTERHEART Latin American study. Circulation. 2007 Mar 6;115(9):1067-74. doi: 10.1161/CIRCULATIONAHA.106.633552. PMID 17339564
- [Background] Lopez-Jaramillo P, Silva SY, Rodriguez-Salamanca N, Duran A, Mosquera W, Castillo V. Are nutrition-induced epigenetic changes the link between socioeconomic pathology and cardiovascular diseases? Am J Ther. 2008 Jul-Aug;15(4):362-72. doi: 10.1097/MJT.0b013e318164bf9c. PMID 18645341
- [Background] Pi-Sunyer FX. The obesity epidemic: pathophysiology and consequences of obesity. Obes Res. 2002 Dec;10 Suppl 2:97S-104S. doi: 10.1038/oby.2002.202. PMID 12490658
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] Ford ES, Giles WH, Dietz WH. Prevalence of the metabolic syndrome among US adults: findings from the third National Health and Nutrition Examination Survey. JAMA. 2002 Jan 16;287(3):356-9. doi: 10.1001/jama.287.3.356. PMID 11790215
- [Background] Perez M, Casas JP, Cubillos-Garzon LA, Serrano NC, Silva F, Morillo CA, Lopez-Jaramillo P. Using waist circumference as a screening tool to identify Colombian subjects at cardiovascular risk. Eur J Cardiovasc Prev Rehabil. 2003 Oct;10(5):328-35. doi: 10.1097/01.hjr.0000095050.46631.6f. PMID 14663294
- [Background] Garcia RG, Perez M, Maas R, Schwedhelm E, Boger RH, Lopez-Jaramillo P. Plasma concentrations of asymmetric dimethylarginine (ADMA) in metabolic syndrome. Int J Cardiol. 2007 Nov 15;122(2):176-8. doi: 10.1016/j.ijcard.2006.11.058. Epub 2007 Jan 16. PMID 17234281
- [Background] Karlsson C, Lindell K, Ottosson M, Sjostrom L, Carlsson B, Carlsson LM. Human adipose tissue expresses angiotensinogen and enzymes required for its conversion to angiotensin II. J Clin Endocrinol Metab. 1998 Nov;83(11):3925-9. doi: 10.1210/jcem.83.11.5276. PMID 9814470
- [Background] Arenas IA, Xu Y, Lopez-Jaramillo P, Davidge ST. Angiotensin II-induced MMP-2 release from endothelial cells is mediated by TNF-alpha. Am J Physiol Cell Physiol. 2004 Apr;286(4):C779-84. doi: 10.1152/ajpcell.00398.2003. Epub 2003 Nov 26. PMID 14644777
- [Background] Lundgren M, Svensson M, Lindmark S, Renstrom F, Ruge T, Eriksson JW. Fat cell enlargement is an independent marker of insulin resistance and 'hyperleptinaemia'. Diabetologia. 2007 Mar;50(3):625-33. doi: 10.1007/s00125-006-0572-1. Epub 2007 Jan 10. PMID 17216279
- [Background] Welch C, Wuarin L, Sidell N. Antiproliferative effect of the garlic compound S-allyl cysteine on human neuroblastoma cells in vitro. Cancer Lett. 1992 Apr 30;63(3):211-9. doi: 10.1016/0304-3835(92)90263-u. PMID 1349504
- [Background] Gebhardt R. Inhibition of cholesterol biosynthesis by a water-soluble garlic extract in primary cultures of rat hepatocytes. Arzneimittelforschung. 1991 Aug;41(8):800-4. PMID 1781801
- [Background] Chi MS, Koh ET, Stewart TJ. Effects of garlic on lipid metabolism in rats fed cholesterol or lard. J Nutr. 1982 Feb;112(2):241-8. doi: 10.1093/jn/112.2.241. PMID 7057262
- [Background] Shoetan A, Augusti KT, Joseph PK. Hypolipidemic effects of garlic oil in rats fed ethanol and a high lipid diet. Experientia. 1984 Mar 15;40(3):261-3. doi: 10.1007/BF01947571. PMID 6698185
- [Background] Gebhardt R. Multiple inhibitory effects of garlic extracts on cholesterol biosynthesis in hepatocytes. Lipids. 1993 Jul;28(7):613-9. doi: 10.1007/BF02536055. PMID 8394977
- [Background] Srivastava KC, Tyagi OD. Effects of a garlic-derived principle (ajoene) on aggregation and arachidonic acid metabolism in human blood platelets. Prostaglandins Leukot Essent Fatty Acids. 1993 Aug;49(2):587-95. doi: 10.1016/0952-3278(93)90165-s. PMID 8415808
- [Background] Kiesewetter H, Jung F, Jung EM, Mroweitz C, Koscielny J, Wenzel E. Effect of garlic on platelet aggregation in patients with increased risk of juvenile ischaemic attack. Eur J Clin Pharmacol. 1993;45(4):333-6. doi: 10.1007/BF00265950. PMID 8299665
- [Background] Sendl A, Schliack M, Loser R, Stanislaus F, Wagner H. Inhibition of cholesterol synthesis in vitro by extracts and isolated compounds prepared from garlic and wild garlic. Atherosclerosis. 1992 May;94(1):79-85. doi: 10.1016/0021-9150(92)90190-r. PMID 1632861
- [Background] Amagase H, Petesch BL, Matsuura H, Kasuga S, Itakura Y. Intake of garlic and its bioactive components. J Nutr. 2001 Mar;131(3s):955S-62S. doi: 10.1093/jn/131.3.955S. PMID 11238796
- [Background] Borek C. Antioxidant health effects of aged garlic extract. J Nutr. 2001 Mar;131(3s):1010S-5S. doi: 10.1093/jn/131.3.1010S. PMID 11238807
- [Background] Steiner M, Khan AH, Holbert D, Lin RI. A double-blind crossover study in moderately hypercholesterolemic men that compared the effect of aged garlic extract and placebo administration on blood lipids. Am J Clin Nutr. 1996 Dec;64(6):866-70. doi: 10.1093/ajcn/64.6.866. PMID 8942410
- [Background] Slowing K, Ganado P, Sanz M, Ruiz E, Tejerina T. Study of garlic extracts and fractions on cholesterol plasma levels and vascular reactivity in cholesterol-fed rats. J Nutr. 2001 Mar;131(3s):994S-9S. doi: 10.1093/jn/131.3.994S. PMID 11238804
- [Background] Macan H, Uykimpang R, Alconcel M, Takasu J, Razon R, Amagase H, Niihara Y. Aged garlic extract may be safe for patients on warfarin therapy. J Nutr. 2006 Mar;136(3 Suppl):793S-795S. doi: 10.1093/jn/136.3.793S. PMID 16484565
- [Background] Moncada S, Palmer RM, Higgs EA. Nitric oxide: physiology, pathophysiology, and pharmacology. Pharmacol Rev. 1991 Jun;43(2):109-42. No abstract available. PMID 1852778
- [Background] Palmer RM, Ferrige AG, Moncada S. Nitric oxide release accounts for the biological activity of endothelium-derived relaxing factor. Nature. 1987 Jun 11-17;327(6122):524-6. doi: 10.1038/327524a0. PMID 3495737
- [Background] Kerwin JF Jr, Lancaster JR Jr, Feldman PL. Nitric oxide: a new paradigm for second messengers. J Med Chem. 1995 Oct 27;38(22):4343-62. doi: 10.1021/jm00022a001. No abstract available. PMID 7473563
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Accini JL, Sotomayor A, Trujillo F, Barrera JG, Bautista L, Lopez-Jaramillo P. Colombian study to assess the use of noninvasive determination of endothelium-mediated vasodilatation (CANDEV). Normal values and factors associated. Endothelium. 2001;8(2):157-66. doi: 10.3109/10623320109165324. PMID 11572477
- [Background] Lopez-Jaramillo P, Diaz LA, Pardo A, Parra G, Jaimes H, Chaudhuri G. Estrogen therapy increases plasma concentrations of nitric oxide metabolites in postmenopausal women but increases flow-mediated vasodilation only in younger women. Fertil Steril. 2004 Dec;82(6):1550-5. doi: 10.1016/j.fertnstert.2004.05.083. PMID 15589858
- [Background] Williams MJ, Sutherland WH, McCormick MP, Yeoman DJ, de Jong SA. Aged garlic extract improves endothelial function in men with coronary artery disease. Phytother Res. 2005 Apr;19(4):314-9. doi: 10.1002/ptr.1663. PMID 16041725
- [Background] Garcia RG, Celedon J, Sierra-Laguado J, Alarcon MA, Luengas C, Silva F, Arenas-Mantilla M, Lopez-Jaramillo P. Raised C-reactive protein and impaired flow-mediated vasodilation precede the development of preeclampsia. Am J Hypertens. 2007 Jan;20(1):98-103. doi: 10.1016/j.amjhyper.2006.06.001. PMID 17198919
- [Background] Lopez-Jaramillo P, Herrera E, Garcia RG, Camacho PA, Castillo VR. Inter-relationships between body mass index, C-reactive protein and blood pressure in a Hispanic pediatric population. Am J Hypertens. 2008 May;21(5):527-32. doi: 10.1038/ajh.2007.86. Epub 2008 Mar 6. PMID 18437144
- [Background] Teran E, Escudero C, Moya W, Flores M, Vallance P, Lopez-Jaramillo P. Elevated C-reactive protein and pro-inflammatory cytokines in Andean women with pre-eclampsia. Int J Gynaecol Obstet. 2001 Dec;75(3):243-9. doi: 10.1016/s0020-7292(01)00499-4. PMID 11728484
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Rotter V, Nagaev I, Smith U. Interleukin-6 (IL-6) induces insulin resistance in 3T3-L1 adipocytes and is, like IL-8 and tumor necrosis factor-alpha, overexpressed in human fat cells from insulin-resistant subjects. J Biol Chem. 2003 Nov 14;278(46):45777-84. doi: 10.1074/jbc.M301977200. Epub 2003 Sep 2. PMID 12952969
- [Background] Yeh YY, Yeh SM. Garlic reduces plasma lipids by inhibiting hepatic cholesterol and triacylglycerol synthesis. Lipids. 1994 Mar;29(3):189-93. doi: 10.1007/BF02536728. PMID 8170288
- [Background] World Health Organization. Deaths from coronary heart disease. The Atlas of Heart Disease and Stroke 2006; Available at: http://www.who.int/cardiovascular_diseases/en/cvd_atlas_14_deathHD.pdf.
- [Background] World Health Organization. Global burden of coronary heart disease. The Atlas of Heart Disease and Stroke 2006; Available at: http://www.who.int/cardiovascular_diseases/en/cvd_atlas_13_coronaryHD.pdf
- [Background] Pineda CA. Síndrome Metabólico: definición, historia, criterios. Colombia Médica. 2008; 39 : 96-106.
- [Background] Rueda-Clausen C, Bolivar IC, Calderon J, Fernandez-Alfonso MS, Carreño M, Cachofeiro V, et al. Abdominal obesity is related with changes in vascular reactivity of human internal mammary artery independently of other cardiovascular risk factors. Atherosclerosis Sup. 2007; 8:11.
- [Background] ZLATKIS A, ZAK B, BOYLE AJ. A new method for the direct determination of serum cholesterol. J Lab Clin Med. 1953 Mar;41(3):486-92. No abstract available. PMID 13035283
- [Background] Yamasaki T, Li L, Lau B. Garlic compounds protect vascular endothelial cells from hydrogen peroxide-induced oxidant injury. 1993: Phytother. Res. 8: 408-412.
- [Background] Tadi P, Teel RW, Lau B. Anticandidal and anticarcinogenic potentials of garlic.1990: Int. Clin. Nutr. Rev. 10: 423-429.